CLINICAL TRIAL: NCT05960032
Title: A PHASE 1, OPEN-LABEL, SINGLE DOSE STUDY TO INVESTIGATE THE PHARMACOKINETICS, SAFETY AND TOLERABILITY OF ZAVEGEPANT INTRANASAL ADMINISTRATION IN HEALTHY CHINESE ADULT PARTICIPANTS
Brief Title: A Study to Learn About the Study Medicine Called Zavegepant in Healthy Chinese Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C5301009
Record Dates: First submitted 2023-07-16; First posted 2023-07-25 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: Zavegepant; Healthy volunteer

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Zavegepant (Experimental): Participants receiving Zavegepant for the treatment phase of the study
  Interventions: Drug: Zavegepant

INTERVENTIONS:
Drug: Zavegepant — Participants receiving single dose of Zavegepant 10 mg

SUMMARY:
The purpose of this study is to learn about:

* how Zavegepant is changed and removed from the body after taken.
* safety of Zavegepant.
* the extent to which side effects can be tolerated after taking Zavegepant for the possible short-term treatment of migraine.

This study is seeking participants who:

* are healthy Chinese adults and includes participants who are between 18 to 55 years old.
* have body mass index (BMI) of 18 to 30 kg/m^2.
* have a total body weight of:
* equal to or more than 50 kilograms (110 pounds) for males.
* equal to or more than 45 kilograms (99 pounds) for females.
* are non-smoker (no use of tobacco or nicotine products).

All participants in this study will receive Zavegepant by nose, once at the study clinic.

The experiences of the participants receiving the study medicine will be looked at. This will help see if the study medicine is safe.

Participants will take part in this study for around 9 weeks. During this time, participants will have 2 study visits at the study clinic and 1 contact over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese adults and includes participants who are between 18 to 55 years old
* BMI of 18 to 30 kg/m^2; and a total body weight ≥50 kg (110 lb) for males and ≥45 kg (99 lb) for females
* Non-smoker (no use of tobacco or nicotine products).

Exclusion Criteria:

* Evidence or history of clinically significant disease.
* Use of medication other than topical products without significant systemic absorption.
* Previous participantion in a clinical research study or investigational study prior to the first dosing.
* Any clinically significant abnormal laboratory test results or positive test.
* Evidence of organ dysfunction or any clinically significant deviation from normal.
* Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic).
* Standard 12-lead ECG that demonstrates clinically relevant abnormalities.
* Abnormalities in clinical laboratory tests: AST or ALT level > ULN; Total bilirubin level > ULN; ANC or ALC level > ULN.
* Positive urine drug screen, alcohol breath test, or urine cotinine test.
* Positive pregnancy test.
* Positive result for COVID-19.
* History of significant alcohol abuse or drug abuse.
* History of anaphylaxix reaction or a clinically important reaction to any drug.
* Donation of plasma within 30 days prior to dosing. Donation or loss of blood of approximately 400 mL or more within 60 days prior to dosing.
* Inability to be venipunctured and/or tolerate catheter venous access.
* Habitual use of snuff tobacco.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Huashan Hospital,Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5301009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 13 participants were enrolled and 12 participants received 1 dose of study intervention, and all 12 participants completed the study.
Groups:
- Zavegepant IN 10 mg: Zavegepant 10 mg was administered intranasally (IN) on Day 1.
Period: TREATMENT
Arm/Group | Zavegepant IN 10 mg
Started | 12
Received Treatment | 12
Completed | 12
Not Completed | 0
Period: FOLLOW-UP
Arm/Group | Zavegepant IN 10 mg
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who received study treatments were included in baseline analysis population.
Arm/Group | Zavegepant IN 10 mg
Number analyzed (Participants) | 12
Age, Customized [Count of Participants; unit: Participants]
  <18 Years | 0
  18-25 Years | 3
  26-35 Years | 6
  36-45 Years | 3
  >45 Years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 12

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Zavegepant in Plasma Following Single Dose of Zavegepant 10 mg IN
Description: Maximum plasma concentration (Cmax) was measured.
Time Frame: 0 (pre-dose), 5 min, 10 min, 20 min, 30 min, 40 min, 50 min, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 8 hours, 12 hours, 16 hours, 24 hours post dose on Day 1
Population: The analysis population refers to all participants who were dosed and had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Zavegepant IN 10 mg
Number analyzed (Participants) | 12
nanogram per milliliter (ng/mL) | 20.32 (114)

2. Primary Outcome: AUClast of Zavegepant in Plasma Following Single Dose of Zavegepant 10 mg IN
Description: AUClast, area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration (Clast), was measured.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | Zavegepant IN 10 mg
Number analyzed (Participants) | 12
ng*hour/mL | 44.25 (122)

3. Primary Outcome: AUCinf of Zavegepant in Plasma Following Single Dose of Zavegepant 10 mg IN
Description: AUCinf, area under the plasma concentration-time curve from time 0 extrapolated to infinite time, was measured.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Zavegepant IN 10 mg
Number analyzed (Participants) | 10
ng*hr/mL | 53.53 (128)

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention, including untoward findings on physical examinations captured as AEs if any.
Time Frame: Day 1 up to maximum of 35 days post single dose administration
Population: All participants who took study intervention were included in the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant IN 10 mg
Number analyzed (Participants) | 12
Participants
  With all-causality TEAEs | 4
  With treatment-related TEAEs | 3

5. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Time Frame: Day 1 up to maximum of 35 days post single dose administration
Population: All participants who took study intervention were included in the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant IN 10 mg
Number analyzed (Participants) | 12
Participants | 1

6. Secondary Outcome: Number of Participants With Clinically Significant Values of Vital Signs
Time Frame: Day 1 up to maximum of 35 days post single dose administration
Population: All participants who took study intervention were included in the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant IN 10 mg
Number analyzed (Participants) | 12
Participants | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Values of 12-lead ECGs
Time Frame: Day 1 up to maximum of 35 days post single dose administration
Population: All participants who took study intervention were included in the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Zavegepant IN 10 mg
Number analyzed (Participants) | 12
Participants | 0

8. Secondary Outcome: Tmax of Zavegepant in Plasma Following Single Dose of Zavegepant 10 mg IN
Description: Tmax, time to Cmax, was measured.
Time Frame: as for outcome 1
Population: The analysis population refers to all participants who were dosed and had at least 1 of the PK parameters of secondary interest.
Measure: Median (Full Range); unit: hour
Arm/Group | Zavegepant IN 10 mg
Number analyzed (Participants) | 12
hour | 0.584 [0.333 to 1.00]

9. Secondary Outcome: t1/2 of Zavegepant in Plasma Following Single Dose of Zavegepant 10 mg IN
Description: T1/2, terminal half-life, was measured.
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Zavegepant IN 10 mg
Number analyzed (Participants) | 10
hour | 11.00 (1.4929)

10. Secondary Outcome: CL/F of Zavegepant in Plasma Following Single Dose of Zavegepant 10 mg IN
Description: CL/F, apparent clearance, was measured.
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hr
Arm/Group | Zavegepant IN 10 mg
Number analyzed (Participants) | 10
Liter/hr | 186.8 (128)

11. Secondary Outcome: Vz/F of Zavegepant in Plasma Following Single Dose of Zavegepant 10 mg IN
Description: Vz/F, apparent volume of distribution, was measured.
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Zavegepant IN 10 mg
Number analyzed (Participants) | 10
Liter | 2943 (141)

ADVERSE EVENTS:
Time Frame: Day 1 up to maximum of 35 days post single dose administration
Arm/Group | Zavegepant IN 10 mg
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zavegepant IN 10 mg (N=12)
Laryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal mucosal discolouration (Respiratory, thoracic and mediastinal disorders) | 1
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Urticaria papular (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-02-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT05960032/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT05960032/SAP_001.pdf